CLINICAL TRIAL: NCT03226756
Title: A Safety Study of Nivolumab in Patients With Recurrent and/or Metastatic Platinum-refractory Squamous Cell Carcinoma of the Head and Neck (SCCHN)
Brief Title: Nivolumab in Recurrent and/or Metastatic SCCHN
Acronym: TopNIVO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UNICANCER (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UC-0130/1703; 2017-000424-10 (EudraCT Number)
Record Dates: First submitted 2017-07-04; First posted 2017-07-24 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Recurrent and/or Metastatic Platinum-refractory SCCHN
MeSH Terms: interventions — Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nivolumab (Experimental): All patients enrolled in the study will received Nivolumab injections, 3mg/kg IV, every 2 weeks, up to 12 cycles (1 cycle = 28 days).
  Interventions: Drug: Nivolumab Injection

INTERVENTIONS:
Drug: Nivolumab Injection — Nivolumab 3 mg/kg, every 2 weeks

SUMMARY:
Recurrent and/or metastatic Squamous Cell Carcinoma of the Head and Neck (SCCHN) are a common clinical situation and although this group of patients has very heterogeneous disease characteristics, they share a dismal prognosis with a median survival time around 6-11 months and a relatively poor quality of life.

Immunotherapy approaches have recently demonstrated clinical efficacy in more than twenty cancer types, including melanoma, renal cell carcinoma, non-small cell lung cancer (NSCLC) and SCCHN. Nivolumab demonstrated significant overall survival benefit as treatment for recurrent SCCHN in a randomized phase III Study CA209141 conducted on a cohort of 361 patients (240 in the nivolumab arm and 121 in the standard therapy arm), presenting this condition and whose disease had progressed within 6 months after platinum-based chemotherapy. In this study, treatment with nivolumab resulted in significantly longer survival than treatment with standard therapy with a median overall survival of 7.5 months vs 5.1 months (p=0.01).

The main objective of the study is to provide additional insight into the frequency of high-grade AEs related to nivolumab and their outcome, and thus supplement the growing safety database of nivolumab-treated recurrent and/or metastatic squamous cell carcinoma of the head and neck patients.

ELIGIBILITY:
Diagnosis and inclusion criteria

1. Adult men and women ≥18 years.
2. Histologically confirmed recurrent and/or metastatic SCCHN (oral cavity, pharynx, larynx), stage III/IV and not amenable to local therapy with curative intent (surgery or radiation therapy with or without chemotherapy).
3. Patients with Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
4. Documentation of p16-positive or p16-negative disease to determine human papillomavirus (HPV) status of tumor for SCC of the oropharynx.
5. Tumor progression or recurrence after a platinum therapy in the adjuvant (ie with radiation after surgery), primary (ie, with radiation), recurrent, or metastatic setting. In the adjuvant or primary setting, the recurrence must have occurred within 6 months after the last dose of platinum therapy. Clinical progression after platinum therapy is an allowable event for entry and is defined as progression of a lesion at least 10 mm in size that is amenable to caliper measurement (eg superficial skin lesion as per RECIST v1.1) or a lesion that has been visualized and photographically recorded with measurements and shown to have progressed.
6. Measurable disease by CT or MRI per RECIST v1.1.
7. Prior curative radiation therapy must have been completed at least 4 weeks prior to study drug administration. Prior focal palliative radiotherapy must have been completed at least 2 weeks before study drug administration.
8. Immunosuppressive doses of systemic medication, such as steroids or absorbed topical steroids (doses > 10 mg/day prednisone or equivalent) must be discontinued at least 2 weeks before study drug administration.
9. Patients with brain metastases will be eligible if they are: asymptomatic, without edema, not on corticosteroids, have been treated and there is no magnetic resonance imaging (except where contraindicated in which CT scan is acceptable) evidence of progression for at least 4 weeks after treatment is complete.
10. Screening laboratory values must meet the following criteria (using CTCAE v4) and should be obtained within 7 days prior to the first study drug administration :

    1. White blood cell (WBC) ≥2000/μL.
    2. Polynuclear neutrophils ≥1.5 x 10⁹/L.
    3. Platelets ≥75 x 10⁹/L.
    4. Hemoglobin >8.0 g/mL.
    5. Alanine aminotransferase (ALAT)/aspartate transaminase (ASAT) ≤3.0 x upper limit of normal (ULN) in the absence of liver metastases or ≤5 x ULN in the presence of liver metastases.
    6. Total Bilirubin ≤1.5 x ULN (except Gilbert Syndrome : <3.0 mg/dL)
    7. Creatinine clearance ≥40 mL/min (measured or calculated by Cockcroft and Gault formula) or serum creatinine <2.0 x ULN.
11. Calcium levels must be normalized and maintained within normal limits for study entry and on treatment. Medical management of calcium levels is permitted. Note: Normal calcium levels may be based on ionized calcium or adjusted for albumin.
12. Subjects with an initial magnesium <0.5 mmol/L (1.2 mg/dL) may receive corrective magnesium supplementation but should continue to receive either prophylactic weekly infusion of magnesium and/or oral magnesium supplementation (eg, magnesium oxide) at the investigator's discretion.
13. Potentially reproductive patients must agree to use an effective contraceptive method or practice adequate methods of birth control or practice complete abstinence, 14 days before starting study drug and while on treatment, and for at least 31 weeks (≈ 7 months) for males and 23 weeks (≈ 5 months) for females after the last dose of study drug. Azoospermic males and women of childbearing potential who are continuously not heterosexually active are exempt from contraceptive requirements.
14. Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) done within 24 hours prior to the first dosing.
15. Women who are breastfeeding should discontinue nursing prior to the first dose of study drug and until 6 months after the last dose.
16. Provision of signed and dated, written informed consent prior to any study specific procedures, sampling and analyses.
17. Patients with social insurance coverage.

Non-inclusion criteria

1. Histologically confirmed recurrent and/or metastatic carcinoma of the nasopharynx, squamous cell carcinoma of unknown primary, and salivary gland or non-squamous histologies (eg mucosal melanoma) are not allowed.
2. Any serious or uncontrolled medical disorder that, in the opinion of the investigator, may increase the risk associated with study participation or study drug administration, impair the ability of the subject to receive protocol therapy, or interfere with the interpretation of study results.
3. Prior malignancy active within the previous 3 years except for locally curable cancers that have been apparently cured, such as basal or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the prostate, cervix, or breast.
4. Subjects with active, known or suspected autoimmune disease. Subjects with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
5. Subjects with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days prior to first study drug administration. Inhaled or topical steroids and adrenal replacement doses >10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
6. Patients having received prior therapy with anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-CTLA-4 antibody (or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways).
7. Patients receiving anti-cancer therapies must be discontinued at least 2 weeks prior to administration of study drug. Palliative, focal radiation therapy, and immunosuppressive doses of systemic corticosteroids, except replacement organotherapy (hydrocortisone and fludrocortisone), must be discontinued at least 2 weeks before administration of study drug.
8. All toxicities attributed to prior anti-cancer therapy other than alopecia and fatigue must have resolved to grade 1 (NCI CTCAE version 4) or baseline before administration of study drug. Subjects with toxicities attributed to systemic prior anticancer therapy which are not expected to resolve and result in long lasting sequelae, such as neuropathy after platinum based therapy, are permitted to enroll.
9. Patients with positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS).
10. Patients with positive tests for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV RNA) indicating active or chronic infection.
11. Use of non-oncology vaccines containing live virus for prevention of infectious diseases within 4 weeks prior to study drug. The use of the inactivated seasonal influenza vaccine (Fluzone®) is allowed.
12. Known or underlying medical condition (e.g., a condition associated with diarrhea or acute diverticulitis) that, in the investigator's opinion, would make the administration of study drug hazardous to the patient or obscure the interpretation of toxicity determination or adverse events.
13. History of uncontrolled seizures, central nervous system disorders or psychiatric disability judged by the investigator to be clinically significant, precluding informed consent, or interfering with compliance of oral drug intake (if applicable).
14. Unwillingness to give written informed consent, unwillingness to participate, or inability to comply with the protocol for the duration of the study.
15. Individuals deprived of liberty or placed under the authority of a tutor.
16. Treatment with any other investigational agent, or participation in another clinical trial within 28 days, prior to first study drug administration and during the treatment period.
17. Known history or active symptomatic interstitial lung disease.
18. History of organ transplantation or allogeneic stem cells transplantation .
19. Severe infection requiring parenteral antibiotics treatment.
20. Active tuberculosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 351 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Incidence for high-grade (CTCAE v4.0 Grade 3-4-5) adverse events of interest (AEI). AEI are adverse reactions known to be related to nivolumab (i.e. skin, endocrinopathy, gastrointestinal, hepatic, renal, pulmonary, and hypersensitivity adverse events) | Last dose + 100 days
  The rate (and its 95%CI) of patients who report at least one high-grade (Grade 3-4 and Grade 5) adverse events of interest will be provided.

SECONDARY OUTCOMES:
Time to onset of grade 3+ AEI | last dose + 100 days
  The time to onset of grade 3+ AEI will be estimated by Kaplan-Meier product-limit method. Time to onset is calculated from first dosing date to the grade 3+ onset date. If a patient never experienced the given grade 3+ AEI, the patient will be censored at the date of last dose + 100 days (or at the last contact date if it occurs before date of last dose + 100 days.
Time to resolution of grade 3-4 AEI to grade 1 | the time from the date of grade 3-4 until the date of grade 1, assessed up to 36 months.
  Time to resolution of grade 3-4 will be estimated by Kaplan-Meier method among patients who had experienced this type of AEI from the grade 3-4 AEI onset date to date of AEI grade 1. If an AEI is ongoing at the time of analysis, the time to resolution will be censored at the last contact date.
Rate of patients with at least one or more doses of nivolumab delayed (or cancelled) due to AE | Up to 24 months of treatment
  The rate of patients with one or more doses of nivolumab cancelled due to AE will be estimated.
Rate of patients with nivolumab definitely withdrawn due to AE | Up to 24 months of treatment
  The rate of patients with nivolumab definitively withdrawn due to AEs will be estimated.
Rate of Nivolumab-related deaths | Up to 36 months.
  A monitoring of Nivolumab-related deaths is set-up separately in 2 subgroups of the cohort: among patients with ECOG performance status (PS)of 2 and among patients with ECOG performance status of 0 or 1. The monitoring is the same in the two subgroups. We expect that around half of the patients will have performance status of 2.
  In each subgroup, the monitoring of nivolumab-related deaths will start at the occurrence of the second related death in that subgroup.
Rate of patients who received immune modulating medication or hormonal replacement therapy | Last dose + 100 days
  Management of high-grade adverse events will be characterized by measuring percentage of patients who received immune modulating medication, > 10 mg prednisone equivalents, hormonal replacement therapy in all treated patients and in patients who have experience high-grade adverse events of interest.
Duration of all immune modulating medications given for the select event and summary of patients with resolution of AEs after initiating these therapies. | Last dose + 100 days
  The total duration of all immune modulating medications given for the event will be presented by mean, standard deviation, median, minimum and maximum.
Rate of AEI of maximum grade 1-2 | Last dose + 100 days
  The rate of patients with AEI of highest grade 1-2 during the observation period will be provided.
Overall survival (OS) | Up to 36 months.
  Overall survival is defined as the time from date of inclusion to date of death due to any cause. Patients last known to be alive will be censored at date of last contact. Overall survival will be estimated by Kaplan Meier method.
Progression free survival (PFS) | Up to 36 months.
  Progression-free survival is defined as the time since the inclusion in the trial to the first event among progression and death, whatever the cause of death. Progression is defined according to RECIST 1.1. Patients last known to be alive without progression having occurred before will be censored at date of last contact. Progression free survival will be estimated by Kaplan Meier method.
Objective response rate (ORR) (complete response and partial response according to RECIST 1.1 and to iRECIST) during nivolumab treatment | The time between the fist dose of treatment until the best response, assessed up to 36 months.
  The rate of patients with objective response (complete response or partial response) will be provided. The response is the best response obtained at the evaluations performed during treatment and at the end of treatment. Two evaluations of the response will be done: one according to the RECIST 1.1 criteria and one according the Immune-related Response Criteria (iRECIST).
Pseudo progression | The time between the first dose of treatment until the first confirmed progression, assessed up to 36 months.
  Pseudo-progressions will be described (rate, time of occurrence). Pseudo-progression is defined as a progression according to RECIST 1.1 under treatment (≥ 20% increase in the sum of diameters of target lesions or unequivocal progression of existing non target lesions or new lesion) that is not confirmed, as per iRECIST, at the next evaluation done 4 to 6 weeks later.

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Even, MD, Principal Investigator — Gustave Roussy Cancer Campus - Villejuif
Locations (18):
- France (18):
  - Institut de Cancérologie de l'Ouest, Angers
  - CHU Bordeaux, Bordeaux
  - Centre Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges Francois Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - ICM Val d'Aurelle, Montpellier
  - Centre Antoine Lacassagne, Nice
  - Hopital Tenon, Paris
  - Institut Curie, Paris
  - Institut Jean Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - Institut Curie Saint Cloud, Saint-Cloud
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No